CLINICAL TRIAL: NCT04302337
Title: Comparison of Short and Long-term Results of Conventional Curettage Adenoidectomy Without Endoscopy Assistance Versus Curettage Adenoidectomy With Transoral Endoscopic Residue Ablation in Children
Brief Title: Conventional Curettage Adenoidectomy vs Curettage Adenoidectomy With Transoral Endoscopic Residue Ablation in Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: technical and funding issues
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, BELDAN POLAT, Associate Professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019/1553
Record Dates: First submitted 2020-02-23; First posted 2020-03-10 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Adenoid Hypertrophy
Keywords: adenoidectomy; adenoids; curettage

STUDY DESIGN:
Intervention Model Description: One group will receive conventional cold curettage adenoidectomy treatment while the other group will receive curettage adenoidectomy with transoral endoscopic residue ablation treatment. The patients operated on Tuesdays and Fridays will receive the first treatment while on Mondays and Thursdays the second treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patients are not going to be given the detail about the days, so that they would not know which group they would be in. Care provider and investigator would not know which patient is going to be operated on which day. Outcome assessor would not know which patient received which treatment while examining for the long term results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Conventional Curettage Adenoidectomy (Active Comparator): Adenoidectomy with Beckmann Adenoid Curette
  Interventions: Procedure: Conventional cold curettage adenoidectomy
- Curettage Adenoidectomy With Transoral Endoscopic Ablation (Experimental): Transoral endoscopic adenoidectomy with Coblator 2 system
  Interventions: Procedure: Curettage adenoidectomy with transoral endoscopic ablation

INTERVENTIONS:
Procedure: Curettage adenoidectomy with transoral endoscopic ablation — Transoral endoscopic examination of nasopharynx at the end of cold curettage adenoidectomy, and, if found, ablation of residual tissue.
  Arms: Curettage Adenoidectomy With Transoral Endoscopic Ablation
Procedure: Conventional cold curettage adenoidectomy — Conventional cold curettage adenoidectomy without endoscopic examination for residual tissue.
  Arms: Conventional Curettage Adenoidectomy

SUMMARY:
This prospective study is designed to compare short and long term results of conventional cold curettage adenoidectomy in children performed without doing any endoscopic or mirror examination before ending the operation versus when combined with transoral endoscopic residue ablation using a wand.

DETAILED DESCRIPTION:
Residual or recurrent adenoid tissue that causes persistence or recurrence of symptoms is observed frequently after conventional cold curettage adenoidectomy. New techniques to better visualize or excise the tissue in order to prevent this situation are being developed. This study aims to compare transoral endoscopic controlled adenoidectomy with conventional blind curettage adenoidectomy in terms of recurrent adenoid hypertrophy. Although there are other studies comparing the results of the two techniques in terms of early residual adenoid tissue and bleeding, no studies comparing the long term results were found in literature. This prospective study is planned to focus on both early examination of residual tissue and long term recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients within 3-12 years old
* Patients undergoing tonsillectomy and adenoidectomy for obstructive sleep disorder
* Patients undergoing adenoidectomy and ventilation tube insertion for chronic otitis media with effusion (OME)
* Patients undergoing adenoidectomy alone for obstructive sleep disorder
* Patients undergoing adenoidectomy alone for chronic OME
* Patients undergoing adenoidectomy alone for chronic sinusitis

Exclusion Criteria:

* Patients not between 3-12 years old
* Patients with craniofacial anomalies
* Revision adenoidectomy
* Proven significant comorbidities
* Systemic diseases
* Bleeding diathesis

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Residual adenoid tissue evaluation with Parikh grade | 1 year after surgery
  Endoscopic examination of adenoid tissue postoperatively

SECONDARY OUTCOMES:
Bleeding | Up to 2 weeks after surgery
  The frequency of postoperative bleeding complication
Otitis media with effusion | Up to 1 year after surgery
  Persistency and recurrence of OME after adenoidectomy

CONTACTS AND LOCATIONS:
Overall Officials: Beldan Polat, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bidaye R, Vaid N, Desarda K. Comparative analysis of conventional cold curettage versus endoscopic assisted coblation adenoidectomy. J Laryngol Otol. 2019 Apr;133(4):294-299. doi: 10.1017/S0022215119000227. Epub 2019 Mar 19. PMID 30885281